CLINICAL TRIAL: NCT04099563
Title: A PHASE 1, OPEN-LABEL, SINGLE-ARM, SINGLE DOSE AND MULTIPLE DOSES STUDY TO ASSESS PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF-04965842 IN CHINESE HEALTHY PARTICIPANTS
Brief Title: Study to Assess Pharmacokinetics, Safety and Tolerability of PF-04965842 in Chinese Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7451028
Record Dates: First submitted 2019-09-03; First posted 2019-09-23 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: HEALTHY
MeSH Terms: interventions — abrocitinib; Tablets

STUDY DESIGN:
Intervention Model Description: open-label, single-arm, single- and multiple-dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PF-04965842 (Experimental): Following an overnight fast for at least 10 hours, participants will receive PF-04965842 oral single dose of 200 mg (2 × 100 mg tablets) on Day 1, at approximately 08:00 am plus or minus 2 hours in the morning. On Days 3 to 8, participants will receive PF-04965842 oral dose of 200 mg (2 × 100 mg tablets) QD in the morning at approximately similar clock hour as on Day 1. On Day 3 and Day 6-8, the dosing of PF-04965842 will be after collection of pre-dose blood samples (under fasted condition for at least 10 hours). On Day 8, the dosing will be under fasted condition at approximately 8:00 am plus or minus 2 hours in the morning.
  Interventions: Drug: PF-04965842

INTERVENTIONS:
Drug: PF-04965842 — For this study, the investigational product is PF-04965842 (provided as 100 mg tablet).
  PF-04965842 100 mg tablets will be provided by Pfizer. Investigational product will be presented to the participants in individual dosing containers
  Other Names: Following an overnight fast for at least 10 hours, participants will receive PF-04965842 oral single dose of 200 mg (2 × 100 mg tablets) on Day 1, at approximately 08:00 am plus or; minus 2 hours in the morning, and repeated doses on Day 3 to 8. On Day 8, the dosing will be under fasted; condition at approximately 8:00 am plus or minus 2 hours in the morning.

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, safety and tolerability of PF-04965842 after single dose and once-daily multiple-doses in Chinese healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-arm, single- and multiple-dose study to assess the pharmacokinetics, safety and tolerability of PF-04965842 in Chinese healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 19 to 26 kg/m2; and a total body weight >50 kg.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

* Evidence or clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic (including alcoholic liver disease, nonalcoholic steatohepatitis (NASH), autoimmune hepatitis, and hereditary liver diseases), psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb) and serological reaction of syphilis. As an exception, a positive hepatitis B surface antibody (HBsAb) finding as a result of participant vaccination is permissible.
* Evidence or history of clinically significant dermatological condition (eg, contact dermatitis or psoriasis) or visible rash present during physical examination.
* History of tuberculosis (TB) or active or latent or inadequately treated infection, positive QuantiFERON- TB Gold test or positive chest radiographs for active tuberculosis infection.
* Any history of chronic infections, any history of recurrent infections, any history of latent infections, or any acute infection within 2 weeks of baseline.
* History of disseminated herpes zoster, or disseminated herpes simplex, or recurrent localized dermatomal herpes zoster.
* Have any malignancies or have a history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
* A positive urine drug test.
* Screening sitting blood pressure (BP) >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level >=1.5 × upper limit of normal (ULN); Total bilirubin level >1 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <=1 × ULN.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-11-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | The pharmacokinetic samples will be collected at 0 (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours after dosing on Day 1
  PK parameters derived from plasma PF-04965842 concentration
Maximum Observed Plasma Concentration (Cmax) | The pharmacokinetic samples will be collected at 0 (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours after dosing on Day 1
  PK parameters derived from plasma PF-04965842 concentration
Time to Reach Maximum Observed Plasma Concentration (Tmax) | The pharmacokinetic samples will be collected at 0 (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours after dosing on Day 1
  PK parameters derived from plasma PF-04965842 concentration
Area under the plasma concentration time profile from time zero to time tau | The pharmacokinetic samples will be collected at 0 (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours after dosing on Day 1 and Day8
  PK parameters derived from plasma PF-04965842 concentration

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Screening up to follow up (71 days)
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants With Clinically Significant Change From Baseline in Laboratory Tests | Screening up to follow up (71 days)
  Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Number of Pariticipants With Clinically Significant Change From Baseline in Vital Signs | Screening up to follow up (71 days)
  Sitting BP will be measured with the participant's arm supported at the level of the heart, with feet flat on the floor and back supported, and recorded to the nearest mm Hg after approximately 5 minutes of rest.
Number of Participants With Clinically Significant Treatment-emergent Electrocardiogram (ECG) Findings | Screening up to follow up (71 days)
  All scheduled ECGs should be performed after the participant has rested quietly for at least 10 minutes in a supine position.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Beijing Hospital Sub-Center of Beijing Hospital Clinical Trial & Research Center, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451028